CLINICAL TRIAL: NCT04839406
Title: The Caregiver Pathway - An Intervention to Support Caregivers of Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: The Dam Foundation (Other)
Responsible Party: Principal Investigator, Elin Børøsund, Senior researcher, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 199446
Record Dates: First submitted 2021-03-24; First posted 2021-04-09 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Caregiver Stress Syndrome
Keywords: Caregivers; Post traumatic stress; Health related quality of life; Intensive care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Structured follow up at the ICU
  * 1-3 days after admittance: Map caregivers' prioritized symptoms, needs and preferences with a digital assessment tool, followed by a meeting with a nurse to address these issues.
  * Every 1-2 weeks: Repeat assessment of symptoms and needs with the assessment tool followed by a meeting with a nurse.
  * At discharge: Structured conversation focusing on information and preparation for the transition to a regular ward or to another hospital including a card with information and support.
  * Bereavement: Individualized support based on caregiver expressed needs, preferences and previous mapping, including a card with information and support.
  * Follow up: Caregivers or bereaved will be contacted after 4-6 weeks, and will be offered a follow up conversation either on phone or at the unit.
  Interventions: Behavioral: Structured support of caregivers at the ICU
- Follow up as usual (Control) (No Intervention): Follow up as usual at the ICU

INTERVENTIONS:
Behavioral: Structured support of caregivers at the ICU — Structured support of caregivers at the ICU provided by a trained group of 10-15 ICU nurses
  Arms: Intervention

SUMMARY:
The aim of the project is to test the efficacy of a systematic intervention for individual follow-up of caregivers at the intensive care unit during a 12 month randomized controlled trial.

DETAILED DESCRIPTION:
Caregivers of patients admitted to an intensive care unit (ICU) often experience the situation as traumatic and stressful. Long term consequences such as fatigue, anxiety, depression and symptoms of post-traumatic stress are reported among 30-50 percent of the caregivers of critically ill patients. The need for supportive interventions is called for.

The overall goal of this project is to improve the support for caregivers of intensive care patients. A systematic intervention for individual support of caregivers, The Caregiver Pathway Intervention, has been developed with a multidisciplinary approach, based on existing evidence, through interviews with former caregivers, workshops with health care personnel and user input and testing. The intervention consist of mapping of caregivers' prioritized symptoms, needs and preferences with a digital assessment tool, followed by a meeting with a nurse to address these issues, a structured conversation at discharge, and an invitation to a follow-up conversation 4-6 weeks after discharge/patients death.

The aim of the project is to test the efficacy of The Caregiver Pathway Intervention among caregivers at the ICU in a randomized controlled trial, using outcome measures such as symptoms of post-traumatic stress, anxiety/depression, cost-utility measures and health-related quality of life. The participants will be randomly assigned to The Caregiver Pathway Intervention or the follow-up as usual group. Both groups will receive outcome measures at baseline and at 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of patients admitted to the intensive care unit that is expected to receive invasive mechanical ventilation for at least 48 hours
* Between 18 and 70 years old
* Able to understand and speak Norwegian

Exclusion Criteria:

• None

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Post traumatic stress | Group differences at f-up month 3
  Post traumatic stress will be measured with the Impact of Event Scale-Revised (IES_R). The total score for the IES_R ranges from 0 to 88. A higher score represents more severe symptoms of post traumatic stress disorder.
Post traumatic stress | Group differences at f-up month 6
  Post traumatic stress will be measured with the Impact of Event Scale-Revised (IES_R). The total score for the IES_R ranges from 0 to 88. A higher score represents more severe symptoms of post traumatic stress disorder.
Post traumatic stress | Group differences at f-up month 12
  Post traumatic stress will be measured with the Impact of Event Scale-Revised (IES_R). The total score for the IES_R ranges from 0 to 88. A higher score represents more severe symptoms of post traumatic stress disorder.
Anxiety and Depression | Change from baseline to f-up month 3
  Anxiety and Depression will be measured with the Hospital Anxiety and Depression Scale (HADS). HADS consists of 14 items, and two subscales with seven items respectively. Score range is 0-21 for each subcale.
  Scores: 0-7= Normal, 8-10= Borderline abnormal (borderline case), 11-21= abnormal (case).
Anxiety and Depression | Change from baseline to f-up month 6
  Anxiety and Depression will be measured with the Hospital Anxiety and Depression Scale (HADS). HADS consists of 14 items, and two subscales with seven items respectively. Score range is 0-21 for each subcale.
  Scores: 0-7= Normal, 8-10= Borderline abnormal (borderline case), 11-21= abnormal (case).
Anxiety and Depression | Change from baseline to f-up month 12
  Anxiety and Depression will be measured with the Hospital Anxiety and Depression Scale (HADS). HADS consists of 14 items, and two subscales with seven items respectively. Score range is 0-21 for each subcale.
  Scores: 0-7= Normal, 8-10= Borderline abnormal (borderline case), 11-21= abnormal (case).
Quality Adjusted Life Years (QUALYs) | Group differences at f-up month 12
  Quality Adjusted Life Years (QUALYs), an economic evaluation of the quality and quantity of life lived, will be derived from the RAND-12 (Short form health survey, developed by the non profit RAND corporation). QUALY scores range from 1 (perfect health) to 0 (death).

SECONDARY OUTCOMES:
Health related quality of life | Change from baseline to f-up month 3
  Health related quality of life will be measured with the RAND-12 (short form health survey, developed by the non profit RAND corporation). Units is summary score and sub-scale scores. Score range: 0-100 for all scales. Lower scores indicates more disability (0 = maximum disability, 100 = no disability).
Health related quality of life | Change from baseline to f-up month 6
  Health related quality of life will be measured with the RAND-12 (short form health survey, developed by the non profit RAND corporation). Units is summary score and sub-scale scores. Score range: 0-100 for all scales. Lower scores indicates more disability (0 = maximum disability, 100 = no disability).
Health related quality of life | Change from baseline to f-up month 12
  Health related quality of life will be measured with the RAND-12 (short form health survey, developed by the non profit RAND corporation). Units is summary score and sub-scale scores. Score range: 0-100 for all scales. Lower scores indicates more disability (0 = maximum disability, 100 = no disability).
Hope | Change from baseline to f-up month 3
  Hope will be measured with Herth Hope Index (HHI). The summary score ranges between 12-48, and a higher score indicates a higher level of hope.
Hope | Change from baseline to f-up month 6
  Hope will be measured with Herth Hope Index (HHI). The summary score ranges between 12-48, and a higher score indicates a higher level of hope.
Hope | Change from baseline to f-up month 12
  Hope will be measured with Herth Hope Index (HHI). The summary score ranges between 12-48, and a higher score indicates a higher level of hope.
Self-Efficacy. | Change from baseline to f-up month 3
  Self-efficacy will be measured with the General Self-Efficacy Scale (GSE). The summary score range between 10-40, and a higher score indicates higher perceived self-efficacy.
Self-Efficacy. | Change from baseline to f-up month 6
  Self-efficacy will be measured with the General Self-Efficacy Scale (GSE). The summary score range between 10-40, and a higher score indicates higher perceived self-efficacy.
Self-Efficacy. | Change from baseline to f-up month 12
  Self-efficacy will be measured with the General Self-Efficacy Scale (GSE). The summary score range between 10-40, and a higher score indicates higher perceived self-efficacy.
Caregiver satisfaction. | Group differences at f-up month 3
  Caregiver satisfaction will be mesured with the Family satisfaction in the ICU questionnaire (FS-ICU-24). Score range: 0-100, a higher score indicates more satisfaction.
Caregivers burden | Group differences at f-up month 12
  The Caregiver Reaction Assessment (CRA). Summary score range between 5 and 120. A higher score indicates a higher level of burden.
Complicated grief | Group differences at f-up month 12
  Complicated grief will be measured with the Inventory of Complicated Grief (ICG). Summary score range between 0-76, and a higher score indicates risk of complicated grief.

CONTACTS AND LOCATIONS:
Overall Officials: Elin Børøsund, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watland S, Solberg Nes L, Hanson E, Ekstedt M, Stenberg U, Borosund E. The Caregiver Pathway, a Model for the Systematic and Individualized Follow-up of Family Caregivers at Intensive Care Units: Development Study. JMIR Form Res. 2023 Apr 25;7:e46299. doi: 10.2196/46299. PMID 37097744
- [Result] Watland S, Solberg Nes L, Ekeberg O, Rostrup M, Hanson E, Ekstedt M, Stenberg U, Hagen M, Borosund E. The Caregiver Pathway Intervention Can Contribute to Reduced Post-Intensive Care Syndrome Among Family Caregivers of ICU Survivors: A Randomized Controlled Trial. Crit Care Med. 2025 Mar 1;53(3):e555-e566. doi: 10.1097/CCM.0000000000006546. Epub 2024 Dec 24. PMID 39718436